CLINICAL TRIAL: NCT03127748
Title: Changes in Ventricular Remodeling and Exercise Cardiopulmonary Function After Transcatheter Closure of Ventricular Septal Defect
Brief Title: Cardiac Function After Transcatheter VSD Closure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: E-DA Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201503039RINB
Record Dates: First submitted 2015-06-21; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Ventricular Septal Defect
Keywords: ventricular septal defect,transcatheter closure
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
With advances in interventional cardiac catheterization, ventricular septal defect (VSD) could be successfully treated via transcatheter device closure. Cardiac catheterization team of National Taiwan University Children's Hospital has recently treated more than 60 patients with VSD using this technique. Both treatment effect and follow-up results were encouraging. Of particular notice is that many patients experienced subjective improvement in exercise tolerance after VSD closure. Traditionally, VSD could only be repaired by open-heart surgery under cardiopulmonary bypass. Therefore, VSD closure would be considered only for those with moderate to large defect, significant heart failure, or presenting with significant exercise intolerance. With the success in transcatheter closure of VSD, a procedure which is safer and leading to faster recovery comparing to cardiac surgery, device closure of VSD would be a reasonable and sensible treatment of choice if it is beneficial for long-term cardiac function and exercise performance.

This project will prospectively enroll 50 patients with VSDs subject to transcatheter closure of the defect in our institute. Before device closure and 6 months after closure, participants will be assessed with image studies (including speckle tracking and tissue Doppler echocardiography), measurements of serum biomarkers (including B-type natriuretic peptide and biomarkers of collagen metabolism), and standard cardiopulmonary exercise test. The purpose of this study is to investigate the potential benefits of closing VSD with respect to cardiac function and exercise performance, which might serve as basis to redefine future indication of VSD closure.

DETAILED DESCRIPTION:
The investigators will enroll 50 consecutive patients with VSDs from the outpatient clinic of National Taiwan University Children's Hospital and Yi-Da Hospital. All participants will receive transcatheter VSD closure after comprehensive discussion with the clinical physicians and the performing clinicians. However, the investigators do not assign such treatment to the subjects of the study, and are not involved in treatment decision making. The inclusion criteria included:

1. subject to transcatheter device closure of VSD (mostly using Amplatzer ductal occluder I and II for perimembranous VSD, and Amplatzer muscular VSD occluder for muscular VSD) based on clinical need;
2. age between 12-60 years;

Patients with following conditions will be excluded:

1. additional hemodynamically significant structural anomalies, including more than mild degree of VSD-related aortic regurgitation or right ventricular outflow tract obstruction;
2. pulmonary hypertension documented during cardiac catheterization;
3. musculoskeletal anomalies limiting the performance of exercise testing;
4. taking cardiac medications within 6 months of enrollment;
5. having alcohol abuse, coronary artery disease, systemic hypertension, diabetes mellitus, liver disease, renal insufficiency, metabolic bone disease, autoimmune disease, and received operation or having a history of trauma within 6 months of study enrollment.

All study participants will provide written informed consent, and the institutional review committee approved the study protocol. This study conformed to the principles of the Helsinki Declaration.

Study protocols Participants will receive following paired evaluations both before VSD closure and 6 months after VSD closure.

1. Echocardiography The echocardiographic studies will be performed with a commercially available ultrasonography system (iE33, Philips, Andover, Massachusetts). The size of VSD and diameter of aortic annulus will be recorded. The severity of valvular regurgitation will be carefully assessed using standard criteria.5 Global LV function will be assessed by measuring LV end-systolic and end-diastolic dimensions and the LV ejection fraction using the modified biplane Simpson's rule. E- and A-wave velocity of mitral inflow, E-wave deceleration time, isovolumic relaxation time, and pre-ejection time and ejection of LV will be measured using conventional Doppler echocardiography.

   Pulsed-wave tissue Doppler imaging (TDI) will be recorded at medial and lateral mitral annulus at apical 4-chamber view. Five consecutive beats will be recorded from each view. Global LV strain and strain rate will be assessed with 2D speckle tracking analysis at the apical four-chamber view and parasternal short-axis view (mid-ventricular level). Frame rates ranges from 40 to 100 frames/s. During analysis the endocardial border will be manually traced at end-systole and the region of interest width adjusted to include the entire myocardium. The software then automatically tracks the motion of the region of interest. The tracking will avoid areas with VSD (before closure) and device in situ (after closure). Longitudinal, radial, and circumferential strain/strain rates will be recorded.
2. Cardiopulmonary exercise test (CPX) The symptom-limited exercise test was performed on a cycle ergometer (Corival; Lode BV, Zernikepark 16, Groningen, the Netherland) in an upright position, using a ramp wise increase of load depending on the expected individual physical capacity. Oxygen consumption (VO2), carbon dioxide production (VCO2), and minute ventilation (VE) were measured using a breath-by-breath automatic gas analyzer (Cortex MetaMax 3B system, Leipzig, Germany), and the peak respiratory exchange ratio (RER, defined as the ratio of VCO2 to VO2) was recorded. The peak exercise rating of perceived exertion was measured using the Borg scale of perceived exertion (from 6 to 20).

   To evaluate the peak exercise capacity, present study enrolled only patients who achieved maximal exercise effort, which was defined as a peak RER ≥ 1.10, and whose rating of perceived exertion was at least 15 on the Borg scale 6. The 2 maximal exercise parameters, peak VO2, and heart rate reserve, were evaluated. The technical details of measuring peak VO2 have been published elsewhere 7. Peak VO2 was then expressed as the percentage of the predicted value.8, 9, and a percentage of the predicted peak VO2 ≤ 70% was defined as significant exercise intolerance.10 The heart rate reserve was calculated as the difference between peak and resting heart rates.11 Two submaximal exercise parameters were also evaluated. The relationship between oxygen consumption and ventilation was evaluated according to the oxygen uptake efficiency slope (OUES). This was calculated by performing a linear regression of VO2 on the common logarithm of VE by using the equation VO2 = a log (VE) + b. The slope "a" represents the rate of increase in VO2 in response to an increase in VE, and is the called the OUES,12 which was subsequently expressed as the percentage of predicted values.13 In addition, the VE/VCO2 slope, which represents the relationship between ventilation and carbon dioxide production, was calculated. This parameter was obtained by performing linear regression analysis of the data acquired throughout the entire period of the exercise. 14
3. Measurement of serum biomarkers Venous blood samples will be obtained before CMR study. Serum will be isolated within 30 min of phlebotomy and stored at -80°C prior to simultaneous analysis of biomarkers of collagen metabolism. Serum carboxy-terminal propeptide of procollagen type I (PICP) concentration will be determined by sandwich enzyme immunosorbent assay using the METRA EIA kit (Quidel, San Diego, California, USA), and carboxy-terminal telopeptide of collagen type I (CITP) will be determined using a commercial radioimmunoassay (Orion Diagnostica, Espoo, Finland).15 The PICP:CITP ratio was considered an index of the degree of coupling between the synthesis and degradation of collagen type I.15 Serum levels of MMP-9 and TIMP-1 will be analyzed using commercially available 2-site sandwich enzyme-linked immunosorbent assay (Quantikine R&D Systems, Minneapolis, Minnesota, USA).16 The sera of all subjects will be sent to the measurement of plasma BNP levels utilizing the Biosite Triage BNP test (Biosite, San Diego, Calif).
4. Other investigations Standard 12-lead ECGs will be acquired with a commercially available ECG machine and software (ECGLAB 3.0, powered by DM software Inc., USA, MEIGAOYI Corp). Averaged QRS duration, QT interval, and QTc interval among all 12 leads will be calculated and reviewed by two experienced cardiologists.

General health-related QoL will be assessed by using the shortened Taiwanese version of the QoL questionnaire of the World Health Organization (WHOQOL-BREF-Taiwan), which has been used in adolescents and adults with congenital heart disease previously.17 The following clinical data will be collected from patients' medical records and at the time of clinical evaluations: body weight and height, blood pressure, clinical symptoms and signs suggesting heart failure, New York Heart Association functional class, and hemodynamic data obtained during cardiac catheterization.

Statistical analysis Case number estimation: Based on previous published data in patients with small VSDs, the average peak VO2 is 92% of the predicted, with a standard deviation of 21%. It is assumed that a difference in absolute value of peak VO2 > 20% (i.e., difference > 18.4% of predicted) is not likely attributed to the learning effect. In addition, it is assumed that a standard deviation of difference of 30%. If the alpha value was set at 0.05, and the power at 0.80, then the estimated sample size sufficient to detect meaningful changes in peak VO2 after VSD closure would be 2 × [(1.96 + 0.842)2 × (30%)2] / (18.4%)2 = 42. Therefore, present project would have sufficient case number to explore changes in exercise performance after VSD closure if all cases (n = 50) complete follow-up protocol.

Statistics: Data will be expressed as percentage, mean ± standard deviation, or median (25th-75th percentile), as appropriate. Continuous variables will be analyzed using the two-sample t test or the Mann-Whitney U test, after testing for normality. Categorical variables will be analyzed by the chi-squared test or Fisher's exact test, as appropriate. Paired t-test or Wilcoxon signed-rank test will be used to compare data before and after VSD closure. Potential parameters predicting improvement in exercise performance will be identified using ROC curve analysis. The cut-off values of these predictors will be chosen based on best sum of sensitivity and specificity. All statistical analyses will be performed using the SPSS version 19.0 (SPSS Inc, Chicago, Illinois). A value of p ≤ 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion criteria:

1. subject to transcatheter device closure of VSD (mostly using Amplatzer ductal occluder I and II for perimembranous VSD, and Amplatzer muscular VSD occluder for muscular VSD) based on clinical need;
2. age between 12-60 years

Exclusion criteria:

1. additional hemodynamically significant structural anomalies, including more than mild degree of VSD-related aortic regurgitation or right ventricular outflow tract obstruction;
2. pulmonary hypertension documented during cardiac catheterization;
3. musculoskeletal anomalies limiting the performance of exercise testing;
4. taking cardiac medications within 6 months of enrollment;
5. having alcohol abuse, coronary artery disease, systemic hypertension, diabetes mellitus, liver disease, renal insufficiency, metabolic bone disease, autoimmune disease, and received operation or having a history of trauma within 6 months of study enrollment.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with VSD attempting for transcatheter closure
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in exercise capacity--peak oxygen consumption | 6 months
  Changes in peak VO2 (% of predicted value)
Changes in exercise capacity--heart rate reserve | 6 months
  Changes in heart rate reserve (beats per minute)
Changes in echocardiographic parameters-tissue Doppler imaging | 6 months
  Tissue Doppler derived mitral systolic and diastolic velocities (cm/s)
Changes in echocardiographic parameters-strain and strain rate | 6 months
  2D speckle tracking derived left ventricular longitudinal and circumferential strain (%) and strain rate (1/s)

SECONDARY OUTCOMES:
Changes in serum BNP level | 6 months
  Changes in serum BNP level (pg/mL)
Changes in circulating fibrosis markers | 6 months
  Changes in PICP (ng/mL)
Changes in circulating fibrosis markers | 6 months
  Changes in CITP (ng/mL)
Changes in circulating fibrosis markers | 6 months
  Changes in TIMP-1 (ng/mL)
Changes in circulating fibrosis markers | 6 months
  Changes in MMP-9 (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-An Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chen CA, Wang JK, Lin MT, Chiu HH, Hsu JY, Lin SM, Chang YM, Chiu SN, Lu CW, Wu MH, Yang MC. Exercise Capacity and Ventricular Remodeling After Transcatheter Ventricular Septal Defect Closure in Asymptomatic or Minimally Symptomatic Adolescents and Adults. Circ Cardiovasc Interv. 2020 Jun;13(6):e008813. doi: 10.1161/CIRCINTERVENTIONS.119.008813. Epub 2020 Jun 10. PMID 32519889